CLINICAL TRIAL: NCT02465580
Title: A Phase II Pilot-Study With Low-dose hrIL-2 for the Treatment of Systemic Lupus Erythematosus
Brief Title: A Pilot-Study With Low-dose hrIL-2 for the Treatment of Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Monash University (Other); Beijing ShuangLu Pharmaceutical Co., Ltd. (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Dept. Rheumatology and Immunology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hrIL-2-SLE
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hrIL-2 active (Active Comparator): Intervention：Add hrIL-2 according to the protocol to original treatment. HrIL-2 active: 1 million U doses of human recombinant interleukin-2 s.c. injection
  Interventions: Drug: hrIL-2 active
- hrIL-2 placebo (Placebo Comparator): 1 million U doses of placebo s.c. injection
  Interventions: Drug: hrIL-2 placebo

INTERVENTIONS:
Drug: hrIL-2 active — active group: placebo group =1:1
  Other Names: Human recombinant IL-2
  Arms: hrIL-2 active
Drug: hrIL-2 placebo — active group: placebo group =1:1
  Arms: hrIL-2 placebo

SUMMARY:
Dysfunction of regulatory T (Treg) cells has been detected in diverse autoimmune diseases, which can be promoted by interleukin-2 (IL-2). In a previous small sample trail performed by the investigator's group, the investigators found that the Low-dose IL-2 was effective and well tolerated in active SLE, and the effect was associated with selective modulation of CD4+ T cell subsets.

This clinical study will confirm the efficacy and safety of low dose IL-2 treatment in SLE.

The investigators perform a single-centre, double-blind pilot trial with hrIL-2 in SLE.The investigators evaluate the effectiveness and safeness of low-dose hrIL-2 for Systemic lupus erythematosus by randomized controlled study (hrIL-2 (N = 30) versus placebo group (N = 30)).

DETAILED DESCRIPTION:
Each SLE patients (n=60) with Scores>=8 on SLEDAI received low-dose IL-2 or placebo (active group: placebo group =1:1, 1 million units every other day subcutaneously (HrIL-2 1X 106, ip, Qod) for a period of 14 days. After a 14-day rest, another cycle started) for 3 cycles. The end points were safety and clinical and immunologic response.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology criteria for the diagnosis of SLE，1997.
* Under standard treatment (≥ 2 months) at the time of inclusion
* Background treatment failed to control flares or to permit prednisone tapering
* With at least one of the following manifestations: thrombocytopenia, disease-associated rash, mouth ulcer, non-infectious type of fever, active vasculitis, renal disorder(proteinuria>0.5g/day), neuropsychiatric SLE.
* Positive for at least one of the following laboratory tests: ANA>1:160, anti-dsDNA, immunoglobulin>20g/L, decreased C3 or C4, leukopenia<3×10^9/L, thrombocytopenia<100×10^9/L;
* SLE disease activity index(SLEDAI) ≥ 8.
* Negative HIV test.
* Negative for hepatitis B and C virus.
* Negative urine pregnancy test.
* Written informed consent form.

Exclusion Criteria:

* Sever chronic liver, kidney, lung or heart dysfunction; (heart failure (≥ grade III NYHA), hepatic insufficiency (transaminases> 3N) )
* Serious infection such as bacteremia, sepsis;
* Cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or Basocellular carcinoma);
* High-dose steroid pulse therapy (>1.5mg/kg) or IV bolus of corticosteroids in the last 2 months.
* History of administration of rituximab or other biologics;
* Purified protein derivative (tuberculin) >10mm
* Mental disorder or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give information;
* Inability to comply with IL-2 treatment regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Were SLE Responders (SRI) | week 24
  SRI response was defined as (1) a ≥ 4-point reduction in SELENA-SLEDAI score, (2) no new BILAG A score or ≤ 1 new BILAG B score, and (3) no deterioration from baseline in the physician's global assessment by ≥ 0.3 points.
Evaluation of the safety (type and number of adverse events and serious adverse events) of low-doseIL-2 in patients with SLE | 24 weeks
  Adverse events includes injection site reactions, influenza-like symptoms, infection, fever, tumor, cardiovascular event，drug-induced liver and kidney damage.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD, Principal Investigator — Peking University Institute of Rheumatology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Miao M, Xiao X, Tian J, Zhufeng Y, Feng R, Zhang R, Chen J, Zhang X, Huang B, Jin Y, Sun X, He J, Li Z. Therapeutic potential of targeting Tfr/Tfh cell balance by low-dose-IL-2 in active SLE: a post hoc analysis from a double-blind RCT study. Arthritis Res Ther. 2021 Jun 11;23(1):167. doi: 10.1186/s13075-021-02535-6. PMID 34116715
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] He J, Zhang R, Shao M, Zhao X, Miao M, Chen J, Liu J, Zhang X, Zhang X, Jin Y, Wang Y, Zhang S, Zhu L, Jacob A, Jia R, You X, Li X, Li C, Zhou Y, Yang Y, Ye H, Liu Y, Su Y, Shen N, Alexander J, Guo J, Ambrus J, Lin X, Yu D, Sun X, Li Z. Efficacy and safety of low-dose IL-2 in the treatment of systemic lupus erythematosus: a randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2020 Jan;79(1):141-149. doi: 10.1136/annrheumdis-2019-215396. Epub 2019 Sep 19. PMID 31537547